CLINICAL TRIAL: NCT03927274
Title: A Study of Intratumorally-Administered Topotecan Using Convection-Enhanced Delivery (CED) in Patients With Suspected Recurrent/Progressive World Health Organization (WHO) Grade III or IV (High Grade) Glioma Undergoing Stereotactic Biopsy
Brief Title: Intratumorally-Administered Topotecan Using Convection-Enhanced Delivery in Patients With Grade III/ IV Glioma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19970
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Glioma of Brain
Keywords: Glioma; Brain Tumor; High Grade Glioma
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cleveland Multiport Catheter (CMC) + Topotecan (Experimental): For predominantly enhanced tumors with volume of 8 cc or less, only 1 Cleveland Multiport Catheter (CMC) will be placed and convection-enhanced delivery (CED) will be performed over a 4-hour period within an MRI scanner, with the goal of complete tumor coverage (as evidenced by tracer distribution on MRI). The initial rate will be 1.20 ml/hour (5.0 microliters/minute/microcatheter) and infusion will be monitored by intermittent MRI imaging. The rate may be adjusted upwards during the infusion, in the event of incomplete tumor coverage, or downwards, if new mass effect is apparent. Following completion of the 4-hour infusion, the CMC will be removed. The initial rate for each subsequent patient may be adjusted upwards in increments of up to 5 microliters/minute/microcatheter based upon the tumor coverage and safety characteristics of the previously treated patients.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Topotecan — Intratumorally-administered topotecan using convection-enhanced delivery (CED) in patients with suspected recurrent/progressive High Grade Glioma (HGG) requiring stereotactic biopsy and is focused on investigating topotecan brain tissue distribution and determining the safety, toxicity, and tolerability of intratumorally-administered topotecan.

SUMMARY:
The purpose of this study is to determine if treatment with Topotecan by an alternative method, delivering topotecan directly into brain tumors, is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of supratentorial WHO Grade III or IV Glioma (High Grade Glioma) that has undergone surgical biopsy or resection followed by adjuvant chemoradiotherapy, that has evidence of recurrence or progression based on imaging studies and a stereotactic biopsy is indicated for confirmation of recurrence/progression.
* 18 years of age or older
* Karnofsky Performance Status 70-100;
* MRI demonstration of a stereotactically accessible enhancing or predominantly non- enhancing mass that does not require resection to relieve clinically significant mass effect;
* Participant understands the procedures and agrees to comply with the study requirements by providing written informed consent
* Adequate organ function as indicated in protocol

Exclusion Criteria:

* Participant is mentally or legally incapacitated at the time of the study;
* Known HIV(+) or has been diagnosed with AIDS
* Participation in another investigational drug study in the prior 4 weeks
* Positive pregnancy test in a female
* Patient, in the opinion of the investigator, is likely to be poorly compliant.
* Diffuse subependymal or Cerebral Spinal Fluid (CSF) disease
* Tumors involving the cerebellum
* Tumor enhancement involving both hemispheres
* Active infection requiring treatment
* Unexplained febrile illness
* Radiation or chemotherapy within 4 weeks of enrollment
* Systemic diseases associated with unacceptable anesthesia or operative risk
* Inability to undergo magnetic resonance imaging (MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Distribution of topotecan in tumor tissue | Treatment day 1
  The spatial distribution of intratumorally-administered topotecan will be determined using a gadolinium-based contrast agent, volumetric magnetic resonance imaging, and three-dimensional image reconstruction.

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) experienced by participants | Up to 48 weeks
Extent of topotecan backflow | Treatment day 1
  Investigate the extent to which backflow may be observed on MRI during CED-mediated delivery of topotecan

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vogelbaum, M.D, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://moffitt.org